CLINICAL TRIAL: NCT06815211
Title: A Prospective Study for Real-world Evaluation of the Novel European Academy for Allergy and Clinical Immunology (EAACI) Criteria for Disease Control, Remission and Cure in CRSwNP Utilizing the German National CRS Registry (GENRE CRS)
Brief Title: The German National CRS Registry (GenreCRS): Clinical Evaluation of the New European Academy for Allergy and Clinical Immunology (EAACI) Criteria for CRSwNP Disease Control, Remission and Cure in a Real-World Evidence Study Approach
Acronym: GenreCRS
Status: Not yet recruiting | Type: Observational
Sponsor: Ärzteverband Deutscher Allergologen e.V. (Other)
Collaborators: German Society of Otorhinolaryngology, Head and Neck Surgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: GenreCRS_2024_V1.0
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Chronic Rhinosinusitis (CRS); Chronic Rhinosinusitis (CRS) With and Without Nasal Polyps
Keywords: CRSwNP; CRSsNP; Nasal Polyps; Registry; Patient Reported Outcome Measures (PROM)
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- sinus surgery: all patients who received sinus surgery during the observation period
- biologic treatment: all patients who are treated with a biologic drug
- non-biologic, non-surgery: all patients without surgery or biologic treatment during observation period

SUMMARY:
The objective of the study is to establish a registry of patients diagnosed with Chronic Rhinosinusitis with and without Nasal Polyps (CRSwNP/CRSsNP) to collect comprehensive longitudinal real-world evidence from specialised treatment centres in Germany. The primary analysis will concentrate on the treatment efficacy and safety of biologic drugs with a focus on defining disease Control, Remission, and Cure as well as to validate the corresponding clinical evaluation criteria.

DETAILED DESCRIPTION:
The German national CRS registry (Genre CRS) is a nationwide registry for patients with CRSsNP and CRSwNP that aims to include more than 250 centres in Germany. Genre CRS is operated by the German Societies of Allergology (AeDA) and Otorhinolaryngology (DGHNO) and is based on most advanced digital health technologies, including a wide variety of collected parameters. Additionally, patient-reported outcome measures will be captured via a smart phone app and submitted directly to the registry database. This registry is the first of its kind in Germany. It will be the foundation for answering many critical/pivotal research questions that depend on high quality, extensive longitudinal data provided by the registry for future studies.

One important field of application will be the long-term assessment of RWE on therapeutic antibodies, also known as "biologics". Biologics are a novel treatment option for patients with severe CRSwNP and have led to tremendous treatment success. Chronically ill patients with a long history of severe symptoms and impaired quality of life can now experience a significant improvement in CRSwNP symptoms when treated with a biologic, which has prompted the discussion about disease Control, Remission, and even Cure. So far, internationally accepted and clinically evaluated definitions of these terms are lacking, but would greatly assist clinicians in developing therapeutic strategies, particularly for the long-term management of chronically affected patients. The criteria currently in use, although generally accepted, are not evidence-based and do not reflect the perspectives of patients and healthcare providers. An international expert working group of the European Academy for Allergy and Clinical Immunology (EAACI) has therefore developed such criteria, which now need to be clinically evaluated and validated using the comprehensive longitudinal data from Genre CRS.

Data collection includes a variety of parameters involved in the treatment with biologics, analysis of their long-term efficacy and safety including but not limited to:

* Polyp Size
* SNOT22
* Visual analog scales for nasal congestion, rhinorrhea, pressure/facial pain, sense of smell
* Olfactory function
* Necessity for rescue treatment (sinus surgery, OCS)
* Parameters of co-morbid diseases
* Type 2 biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 12 years
* Patients who are diagnosed with CRS according to internationally valid guidelines (EPOS 2020)
* Patients who provide written informed consent or by a legal representative

Exclusion Criteria:

* Patients below the age of 12 years at initiation
* Patients who do not provide written consent or withdraw their consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients above the age of 18 years of any gender with the diagnosis of CRSwNP and CRSsNP treated by a specialized treatment centre in Germany that is part of the German CRS registry network will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score | 1 year
  Size of nasal polyps from 0-4 per side, with 0=no polyps to 4=large polyps reaching the bottom of the nasal cavity
University of Pennsylvania Smell Identification Test (UPSIT) | 1 year
  smell identification test, 0-40 points, with 0 being the lowest smell function and 40 an excellent smell function
Sniffin' Sticks Identification Test 12 | 1 year
  Smell identification test with 12 items, range 0-12, the higher the score, the better the smell function (0=anosmia, 12=normosmia)
Sniffin' Sticks Identification Test 16 | 1 year
  Smell identification test with 16 items, range 0-12, the higher the score, the better the smell function (0=anosmia, 12=normosmia)
Sinonasal Outcome Test 22 (SNOT22) | 1 year
  quality of life questionnaire with 22 items (score 0-22). 0=no impairment, 22=maximum impairment in all categories
Rescue Treatment | 1 year
  Number of courses of systemic corticosteroids and number of sinus surgeries necessary due to poor treatmentcontrol or exacerbation of CRS-symptoms

SECONDARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | 1 year
  measured in l/min
Blood eosinophils | 1 year
  1/µl
Lund-Mackay Score | 1 year
  opacification of nasal sinuses in CT imaging: scores 0-24 with 0=no opacification and 24 complete opacification of all sinuses
Allergic Rhinitis Visual Analogue Scale (AR-VAS) | 1 year
  symptom severity of allergic rhinitis on a visual analogue scale with 0=no symptoms to 10=worst symptoms imaginable
Forced Expiratory Volume in 1 Second (FEV1) | 1 year
  lung function measured in l
Fractional exhaled nitric oxide (FeNO) | 1 year
  measured in ppb
Immunoglobulin E (IgE) | 1 year
  kU/l

IPD SHARING:
Plan to Share IPD: Undecided